CLINICAL TRIAL: NCT01564537
Title: A Phase 3, Randomized, Double-Blind, Multicenter Study Comparing Oral Ixazomib (MLN9708) Plus Lenalidomide and Dexamethasone Versus Placebo Plus Lenalidomide and Dexamethasone in Adult Patients With Relapsed and/or Refractory Multiple Myeloma
Brief Title: A Phase 3 Study Comparing Oral Ixazomib Plus Lenalidomide and Dexamethasone Versus Placebo Plus Lenalidomide and Dexamethasone in Adult Participants With Relapsed and/or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C16010; 2011-005496-17 (EudraCT Number); CTR20130908 (Registry Identifier: SFDA CTR); U1111-1164-7646 (Registry Identifier: WHO); NL40132.018.12 (Registry Identifier: CCMO); 12/LO/0949 (Registry Identifier: NRES); JapicCTI-132345 (Registry Identifier: JapicCTI); 1015042370 (Registry Identifier: TCTIN); C16010CTIL (Registry Identifier: Israel)
Record Dates: First submitted 2012-03-22; First posted 2012-03-28 (Estimated); Results first posted 2016-01-27 (Estimated); Last update posted 2023-03-10 (Actual); Status verified 2023-02

CONDITIONS: Relapsed Multiple Myeloma; Refractory Multiple Myeloma
Keywords: Drug therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ixazomib + Lenalidomide + Dexamethasone (Experimental): Ixazomib 4 mg, capsules, orally, once, on Days 1, 8 and 15; plus lenalidomide 25 mg, orally, once, on Days 1 through 21; and dexamethasone 40 mg, orally, once, on Days 1, 8, 15 and 22 of a 28-day cycle for multiple cycles until progressive disease (PD) or unacceptable toxicity, whichever occurred first up to end of treatment (EOT) up to approximately 42.9 months.
  Interventions: Drug: Ixazomib; Drug: Lenalidomide; Drug: Dexamethasone
- Placebo + Lenalidomide + Dexamethasone (Placebo Comparator): Ixazomib placebo-matching capsules, orally, once, on Days 1, 8 and 15; plus lenalidomide 25 mg, orally, once, on Days 1 through 21; and dexamethasone 40 mg, orally, once, on Days 1, 8, 15 and 22 of a 28-day cycle for multiple cycles until PD or unacceptable toxicity, whichever occurred first up to approximately 41 months.
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone; Drug: Placebo

INTERVENTIONS:
Drug: Ixazomib — Ixazomib capsules
  Other Names: MLN9708; NINLARO®
  Arms: Ixazomib + Lenalidomide + Dexamethasone
Drug: Lenalidomide — Lenalidomide capsules
Drug: Dexamethasone — Dexamethasone tablets
Drug: Placebo — Ixazomib placebo-matching capsules
  Arms: Placebo + Lenalidomide + Dexamethasone

SUMMARY:
The purpose of this study is to determine whether the addition of oral ixazomib to the background therapy of lenalidomide and dexamethasone improves progression free survival (PFS) in participants with relapsed and/or refractory multiple myeloma (RRMM).

DETAILED DESCRIPTION:
The drug being tested in this study is called Ixazomib. Ixazomib is being tested to treat people who have relapsed and/or refractory multiple myeloma (RRMM). This study will look at progression free survival (PFS), overall survival (OS) and safety in participants who take ixazomib in addition to lenalidomide and dexamethasone compared to placebo in addition to lenalidomide and dexamethasone.

The study enrolled 722 patients. Participants were randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* Ixazomib 4 mg + lenalidomide + dexamethasone
* Placebo (dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient + lenalidomide + dexamethasone

All participants will receive treatment in 28 day cycles until disease progression or unacceptable toxicity.

This multi-center trial will be conducted worldwide. The overall time to participate in this study is approximately 80 months. Participants will make multiple visits to the clinic, and will be contacted every 4 weeks for PFS and every 12 weeks for OS.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants 18 years of age or older.
2. Multiple myeloma diagnosed according to standard criteria either currently or at the time of initial diagnosis.

   NOTE: The initial diagnosis must have been symptomatic multiple myeloma, although the relapsed disease did not need to be symptomatic.
3. Must have had measurable disease, defined by at least 1 of the following 3 measurements:

   * Serum M-protein ≥ 1 g/dL (≥ 10 g/L).
   * Urine M-protein ≥ 200 mg/24 hours.
   * Serum free light chain (FLC) assay: involved FLC level ≥ 10 mg/dL (≥ 100 mg/L), provided that the serum FLC ratio was abnormal.
4. Participants with relapsed and/or refractory multiple myeloma (RRMM) who had received 1 to 3 prior therapies.

   NOTE: population included the following 3 categories of participants:
   * Participants who relapsed from their previous treatment(s) but were not refractory to any previous treatment.
   * Participants who were refractory to all lines of previous treatment(s) (ie, participants who had never responded to any therapies received).
   * Participants who relapsed from at least 1 previous treatment AND additionally were refractory to at least 1 previous treatment. For the purposes of this study, refractory disease was defined as disease progression on treatment or progression within 60 days after the last dose of a given therapy.

   A line of therapy was defined as 1 or more cycles of a planned treatment program. This may have consisted of 1 or more planned cycles of single-agent therapy or combination therapy, as well as a sequence of treatments administered in a planned manner. For example, a planned treatment approach of induction therapy followed by autologous stem cell transplantation, followed by maintenance was considered 1 line of therapy. Autologous and allogenic transplants were permitted.
5. Must have met the following clinical laboratory criteria:

   * Absolute neutrophil count (ANC) ≥ 1000/mm^3 and platelet count ≥ 75,000/mm^3. Platelet transfusions to help participants meet eligibility criteria were not allowed within 3 days prior to randomization.
   * Total bilirubin ≤ 1.5 x the upper limit of the normal range (ULN).
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN.
   * Calculated creatinine clearance ≥ 30 mL/min NOTE: Participants with a low creatinine clearance ≤ 60 mL/min (or ≤ 50 mL/min, according to lenalidomide prescribing information/local practice) were to receive a reduced lenalidomide dose of 10 mg once daily (QD) on Days 1 through 21 of a 28-day cycle. The lenalidomide dose may have been escalated to 15 mg QD after 2 cycles if the participant was not responding to treatment and was tolerating the treatment. If renal function normalized (ie, creatinine clearance >60 mL/min or >50 mL/min, according to lenalidomide prescribing information/local practice) and the participant continued to tolerate this treatment, lenalidomide may then have been escalated to 25 mg QD.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
7. Participants who received prior allogenic transplant must have had no active graft-versus-host disease.
8. Female participants who:

   * Were postmenopausal for at least 24 months before the screening visit, OR
   * Were surgically sterile, OR
   * If they were of childbearing potential must have: had a negative pregnancy test with a sensitivity of at least 25 mIU/mL within 10 to 14 days and again within 24 hours prior to starting Cycle 1 of lenalidomide; either agreed to practice true abstinence, when this was in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal were not acceptable methods of contraception.) OR begun 2 reliable methods of birth control (1 highly effective method and 1 additional effective method) at the same time, at least 28 days before starting study treatment through 90 days after the last dose of study treatment; and agreed to ongoing pregnancy testing AND must have also adhered to the guidelines of the RevAssist program (US participants), RevAid program (Canadian participants), iAccess program (Australian participants), RevMate program (Japanese participants) or The Lenalidomide Pregnancy Risk Minimisation Plan as outlined in the Study Manual (all other participants who were not using commercial supplies).

   Male patients, even if surgically sterilized (ie, status postvasectomy), who:
   * Agreed to practice true abstinence, when this was in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal were not acceptable methods of contraception.) OR
   * Agreed to practice effective barrier contraception during the entire study treatment period and 90 days after the last dose of study treatment if their partner was of childbearing potential, even if they had a successful vasectomy, AND
   * Must have also adhered to the guidelines of the RevAssist program (US participants), RevAid program (Canadian participants), iAccess program (Australian participants), RevMate program (Japanese participants) or The Lenalidomide Pregnancy Risk Minimisation Plan as outlined in the study Manual (all other participants who were not using commercial supplies)
9. Must have been able to take concurrent aspirin 81 to 325 mg daily (or enoxaparin 40 mg subcutaneously daily [or its equivalent] if allergic to aspirin), per published standard or institutional standard of care, as prophylactic anticoagulation.

   NOTE: For participants with prior history of deep vein thrombosis (DVT), low-molecular-weight heparin (LMWH) was mandatory.
10. Voluntary written consent must have been given before performance of any study related procedure not part of standard medical care, with the understanding that consent may have been withdrawn by the participant at any time without prejudice to future medical care.
11. Was willing and able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Was refractory to lenalidomide or proteasome inhibitor-based therapy at any line.

   NOTE: Refractory disease was defined as disease progression on treatment or progression within 60 days after the last dose of a given therapy. Participants who progressed after 60 days from the last dose of a given therapy were considered relapsed and were eligible for inclusion in the study.

   Participants who were refractory to thalidomide-based therapy were eligible.
2. Female participants who were breast feeding or pregnant.
3. Failure to have fully recovered (ie, Grade 1 toxicity) from the effects of prior chemotherapy (except for alopecia) regardless of the interval since last treatment.
4. Major surgery within 14 days before randomization.
5. Radiotherapy within 14 days before randomization.
6. Central nervous system involvement.
7. Infection requiring systemic antibiotic therapy or other serious infection within 14 days before randomization.
8. Diagnosis of Waldenstrom's macroglobulinemia, polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes (POEMS) syndrome, plasma cell leukemia, primary amyloidosis, myelodysplastic syndrome, or myeloproliferative syndrome.
9. Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within 6 months before randomization in the study.
10. Systemic treatment with strong inhibitors of cytochrome P450 (CYP) 1A2 (CYP1A2) (fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of CYP3A (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort within 14 days before randomization in the study.
11. Ongoing or active systemic infection, active hepatitis B or C virus infection, or known human immunodeficiency virus positive.
12. Comorbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the participant inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens (eg, peripheral neuropathy that is Grade 1 with pain or Grade 2 or higher of any cause).
13. Psychiatric illness/social situation that would limit compliance with study requirements.
14. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
15. Inability to swallow oral medication, inability or unwillingness to comply with the drug administration requirements, or gastrointestinal condition that could interfere with the oral absorption or tolerance of treatment.
16. Diagnosed or treated for another malignancy within 2 years before randomization or previously diagnosed with another malignancy and any evidence of residual disease. Participants with nonmelanoma skin cancer or carcinoma in situ of any type were not excluded if they had undergone complete resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 722 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2014-10-01 (Actual); Study Completion 2022-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (24):
- United States (18):
  - University of Arkansas Medical Sciences, Little Rock, Arkansas
  - Pacific Cancer Medical Center Inc, Anaheim, California
  - West Contra Costa Healthcare District, Berkeley, California
  - University of Florida, Gainesville, Florida
  - Cancer & Blood Disease Center, Lecanto, Florida
  - Northwest Georgia Oncology Center, Marietta, Georgia
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - Blood and Cancer Clinic, Fayetteville, North Carolina
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - MUSC Hollings Cancer Center, Charleston, South Carolina
  - Fred Hutchinson Cancer Research, Seattle, Washington
  - West Virginia University Hospitals and Clinic, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (6):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Saint John Regional Hospital, Saint John, New Brunswick
  - CHUM Notre-Dame Hospital, Montreal, Quebec
  - MUHC Glen Site Cedars Cancer Centre, Montreal, Quebec

REFERENCES:
- [Derived] Richardson PG, Kumar SK, Masszi T, Grzasko N, Bahlis NJ, Hansson M, Pour L, Sandhu I, Ganly P, Baker BW, Jackson SR, Stoppa AM, Gimsing P, Garderet L, Touzeau C, Buadi FK, Laubach JP, Cavo M, Darif M, Labotka R, Berg D, Moreau P. Final Overall Survival Analysis of the TOURMALINE-MM1 Phase III Trial of Ixazomib, Lenalidomide, and Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma. J Clin Oncol. 2021 Aug 1;39(22):2430-2442. doi: 10.1200/JCO.21.00972. Epub 2021 Jun 11. PMID 34111952
- [Derived] Di Bacco A, Bahlis NJ, Munshi NC, Avet-Loiseau H, Masszi T, Viterbo L, Pour L, Ganly P, Cavo M, Langer C, Kumar SK, Rajkumar SV, Keats JJ, Berg D, Lin J, Li B, Badola S, Shen L, Zhang J, Esseltine DL, Luptakova K, van de Velde H, Richardson PG, Moreau P. c-MYC expression and maturity phenotypes are associated with outcome benefit from addition of ixazomib to lenalidomide-dexamethasone in myeloma. Eur J Haematol. 2020 Jul;105(1):35-46. doi: 10.1111/ejh.13405. Epub 2020 Apr 15. PMID 32145111
- [Derived] Avet-Loiseau H, Bahlis NJ, Chng WJ, Masszi T, Viterbo L, Pour L, Ganly P, Palumbo A, Cavo M, Langer C, Pluta A, Nagler A, Kumar S, Ben-Yehuda D, Rajkumar SV, San-Miguel J, Berg D, Lin J, van de Velde H, Esseltine DL, di Bacco A, Moreau P, Richardson PG. Ixazomib significantly prolongs progression-free survival in high-risk relapsed/refractory myeloma patients. Blood. 2017 Dec 14;130(24):2610-2618. doi: 10.1182/blood-2017-06-791228. Epub 2017 Oct 20. PMID 29054911
- [Derived] Gupta N, Yang H, Hanley MJ, Zhang S, Liu R, Kumar S, Richardson PG, Skacel T, Venkatakrishnan K. Dose and Schedule Selection of the Oral Proteasome Inhibitor Ixazomib in Relapsed/Refractory Multiple Myeloma: Clinical and Model-Based Analyses. Target Oncol. 2017 Oct;12(5):643-654. doi: 10.1007/s11523-017-0524-3. PMID 28803351
- [Derived] Mateos MV, Masszi T, Grzasko N, Hansson M, Sandhu I, Pour L, Viterbo L, Jackson SR, Stoppa AM, Gimsing P, Hamadani M, Borsaru G, Berg D, Lin J, Di Bacco A, van de Velde H, Richardson PG, Moreau P. Impact of prior therapy on the efficacy and safety of oral ixazomib-lenalidomide-dexamethasone vs. placebo-lenalidomide-dexamethasone in patients with relapsed/refractory multiple myeloma in TOURMALINE-MM1. Haematologica. 2017 Oct;102(10):1767-1775. doi: 10.3324/haematol.2017.170118. Epub 2017 Jul 27. PMID 28751562
- [Derived] Hou J, Jin J, Xu Y, Wu D, Ke X, Zhou D, Lu J, Du X, Chen X, Li J, Liu J, Gupta N, Hanley MJ, Li H, Hua Z, Wang B, Zhang X, Wang H, van de Velde H, Richardson PG, Moreau P. Randomized, double-blind, placebo-controlled phase III study of ixazomib plus lenalidomide-dexamethasone in patients with relapsed/refractory multiple myeloma: China Continuation study. J Hematol Oncol. 2017 Jul 6;10(1):137. doi: 10.1186/s13045-017-0501-4. PMID 28683766
- [Derived] Moreau P, Masszi T, Grzasko N, Bahlis NJ, Hansson M, Pour L, Sandhu I, Ganly P, Baker BW, Jackson SR, Stoppa AM, Simpson DR, Gimsing P, Palumbo A, Garderet L, Cavo M, Kumar S, Touzeau C, Buadi FK, Laubach JP, Berg DT, Lin J, Di Bacco A, Hui AM, van de Velde H, Richardson PG; TOURMALINE-MM1 Study Group. Oral Ixazomib, Lenalidomide, and Dexamethasone for Multiple Myeloma. N Engl J Med. 2016 Apr 28;374(17):1621-34. doi: 10.1056/NEJMoa1516282. PMID 27119237
- [Derived] Moreau P, Hulin C, Macro M, Caillot D, Chaleteix C, Roussel M, Garderet L, Royer B, Brechignac S, Tiab M, Puyade M, Escoffre M, Stoppa AM, Facon T, Pegourie B, Chaoui D, Jaccard A, Slama B, Marit G, Laribi K, Godmer P, Luycx O, Eisenmann JC, Allangba O, Dib M, Araujo C, Fontan J, Belhadj K, Wetterwald M, Dorvaux V, Fermand JP, Rodon P, Kolb B, Glaisner S, Malfuson JV, Lenain P, Biron L, Planche L, Caillon H, Avet-Loiseau H, Dejoie T, Attal M. VTD is superior to VCD prior to intensive therapy in multiple myeloma: results of the prospective IFM2013-04 trial. Blood. 2016 May 26;127(21):2569-74. doi: 10.1182/blood-2016-01-693580. Epub 2016 Mar 21. PMID 27002117
- See also: Related Info — https://www.tourmalinetrialmm1.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 187 sites in Australia, Austria, Belgium, Canada, China, Czech Republic, Denmark, France, Germany, Hungary, Israel, Italy, Japan, Republic of Korea, Netherlands, New Zealand, Poland, Portugal, Romania, Russian Federation, Singapore, Spain, Sweden, Turkey, United Kingdom and US from 01 August 2012 to 08 February 2022.
Pre-assignment Details: Participants with a diagnosis of relapsed and/or refractory multiple myeloma were enrolled in 1 of 2 treatment groups: Ixazomib 4 mg or Ixazomib placebo-matching tablets in combination with lenalidomide, and dexamethasone.
Groups:
- Ixazomib+ Lenalidomide + Dexamethasone: Ixazomib 4 mg, capsules, orally, once, on Days 1, 8 and 15; plus lenalidomide 25 mg, orally, once, on Days 1 through 21; and dexamethasone 40 mg, orally, once, on Days 1, 8, 15 and 22 of a 28-day cycle for multiple cycles until progressive disease (PD) or unacceptable toxicity, whichever occurred first up to end of treatment (EOT) (up to approximately 42.9 months).
- Placebo + Lenalidomide + Dexamethasone: Ixazomib placebo-matching capsules, orally, once, on Days 1, 8 and 15; plus lenalidomide 25 mg, orally, once, on Days 1 through 21; and dexamethasone 40 mg, orally, once, on Days 1, 8, 15 and 22 of a 28-day cycle for multiple cycles until PD or unacceptable toxicity, whichever occurred first (up to approximately 41 months).
Period: Overall Study
Arm/Group | Ixazomib+ Lenalidomide + Dexamethasone | Placebo + Lenalidomide + Dexamethasone
Started | 360 | 362
Intent-to-Treat (ITT) Population (ITT population was defined as all randomized participants.) | 360 | 362
Safety Population (Safety population included all randomized participants who received at least 1 dose of any study drug, regardless of their randomized treatment.) | 361 | 359
Response Evaluable Population (Response-Evaluable population included all participants who received at least 1 dose of study drug, had measurable disease at baseline, and at least 1 post-baseline response assessment.) | 345 | 348
Completed | 259 | 263
Not Completed | 101 | 99
Not completed — Site Terminated by Sponsor | 1 | 0
Not completed — Withdrawal by Subject | 12 | 14
Not completed — Lost to Follow-up | 7 | 3
Not completed — Reason not specified | 81 | 82

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population was defined as all randomized participants.
Groups:
- Ixazomib+ Lenalidomide + Dexamethasone: Ixazomib 4 mg, capsules, orally, once, on Days 1, 8 and 15; plus lenalidomide 25 mg, orally, once, on Days 1 through 21; and dexamethasone 40 mg, orally, once, on Days 1, 8, 15 and 22 of a 28-day cycle for multiple cycles until PD or unacceptable toxicity, whichever occurred first up to EOT (up to approximately 42.9 months).
- Total: Total of all reporting groups
Arm/Group | Ixazomib+ Lenalidomide + Dexamethasone | Placebo + Lenalidomide + Dexamethasone | Total
Number analyzed (Participants) | 360 | 362 | 722
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (9.13) | 65.8 (9.70) | 65.7 (9.41)
Age, Customized [Number; unit: participants]
  ≤65 years | 168 | 176 | 344
  >65-≤75 years | 145 | 125 | 270
  >75 years | 47 | 61 | 108
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 153 | 160 | 313
  Male | 207 | 202 | 409
Race/Ethnicity, Customized [Number; unit: participants]
  White | 312 | 303 | 615
  Black or African American | 7 | 6 | 13
  Native Hawaiian/Other Pacific Islander | 2 | 2 | 4
  Asian | 30 | 34 | 64
  American Indian/Alaska native | 0 | 1 | 1
  Other | 4 | 3 | 7
  Not reported | 5 | 13 | 18
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 9 | 12 | 21
  Not Hispanic or Latino | 341 | 333 | 674
  Not Reported | 8 | 15 | 23
  Missing | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  Russian Federation | 21 | 18 | 39
  Singapore | 2 | 4 | 6
  United States | 28 | 23 | 51
  Portugal | 7 | 8 | 15
  Austria | 5 | 4 | 9
  Netherlands | 3 | 6 | 9
  Sweden | 15 | 12 | 27
  China | 3 | 3 | 6
  Korea, Republic of | 4 | 2 | 6
  Poland | 21 | 20 | 41
  France | 36 | 45 | 81
  Romania | 6 | 6 | 12
  Hungary | 18 | 21 | 39
  United Kingdom | 12 | 8 | 20
  Spain | 16 | 14 | 30
  New Zealand | 28 | 39 | 67
  Canada | 19 | 26 | 45
  Czech Republic | 15 | 21 | 36
  Turkey | 4 | 3 | 7
  Belgium | 7 | 7 | 14
  Denmark | 10 | 7 | 17
  Italy | 24 | 15 | 39
  Israel | 19 | 14 | 33
  Australia | 9 | 8 | 17
  Germany | 8 | 7 | 15
  Japan | 20 | 21 | 41
Stratification Factor: Lines of Prior Therapy [Number; unit: participants]
  1 Line | 212 | 213 | 425
  2 or 3 Lines | 148 | 149 | 297
Stratification Factor: Proteasome Inhibitor [Number; unit: participants]
  Exposed | 250 | 253 | 503
  Naïve | 110 | 109 | 219
Stratification Factor: International Staging System (ISS) Stag at Screening [Number; unit: participants] — Stage I: Serum beta2-microglobulin <3.5 mg/L and albumin ≥3.5 g/dL; Stage II: Neither Stage I or III, meaning that either: beta2-microglobulin level ≥3.5 and <5.5 mg/L (with any albumin level), OR albumin <3.5 g/dL with beta2-microglobulin <3.5 mg/L; Stage III: Serum beta2-microglobulin ≥5.5 mg/L. Normal serum beta2-microglobulin: <3.0 mg/L; normal albumin: 3.5-5.0 g/dL.
  participants
    Stage I or Stage II | 314 | 318 | 632
    Stage III | 46 | 44 | 90

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) as Assessed by the Independent Review Committee (IRC)
Description: Progression Free Survival (PFS) is defined as the time from the date of randomization to the date of first documentation of disease progression (PD) or death due to any cause, whichever occurs first. Response including PD was assessed by independent review committee (IRC) using the International Myeloma Working Group (IMWG) response criteria. PD requires 1 of the following: Increase of ≥ 25% from nadir in: Serum M-component (absolute increase ≥ 0.5 g/dl); Urine M-component (absolute increase ≥ 200 mg/24 hours); In patients without measurable serum and urine M-protein levels the difference between involved and uninvolved free light chain (FLC) levels (absolute increase > 10 mg/dl); Development of new or increase in the size of existing bone lesions or soft tissue plasmacytomas; Development of hypercalcemia (corrected serum calcium > 11.5 mg/dl) attributed solely to plasma cell proliferative disease. Status evaluated every 4 weeks until disease progression (PD) was confirmed.
Time Frame: From date of randomization until disease progression or death up to approximately 27 months (approximate median follow-up 15 months)
Population: ITT population was defined as all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib+ Lenalidomide + Dexamethasone | Placebo + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 360 | 362
months | 20.6 [17.02 to NA] — The upper limit of 95% confidence interval was not estimable due to low number of participants with events. | 14.7 [12.91 to 17.58]
Statistical Analysis 1: Comparison: Ixazomib+ Lenalidomide + Dexamethasone vs Placebo + Lenalidomide + Dexamethasone; Test type: Superiority or Other; p = 0.012, Log Rank; Hazard Ratio (HR) = 0.742, 95% CI 2-sided [0.587 to 0.939] — HR is estimated from Cox Regression

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from the date of randomization to the date of death. Participants without documentation of death at the time of the analysis were censored at the date when they were last known to be alive.
Time Frame: From date of randomization until death (up to approximately 97 months)
Population: ITT population was defined as all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib+ Lenalidomide + Dexamethasone | Placebo + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 360 | 362
months | 53.6 [49.25 to 62.95] | 51.6 [44.78 to 59.14]
Statistical Analysis 1: Comparison: Ixazomib+ Lenalidomide + Dexamethasone vs Placebo + Lenalidomide + Dexamethasone; Test type: Superiority; p = 0.495, Log Rank; Hazard Ratio (HR) = 0.939, 95% CI 2-sided [0.784 to 1.125] — HR:estimated from Cox Regression with stratification factors: prior therapies, proteasome inhibitor, and ISS Stage at Screening with treatment as factor in model. <1 hazard ratio for treatment=better prevention of death in drug arm vs control

3. Secondary Outcome: Overall Survival in High-Risk Participants Carrying Deletion 17 [Del(17)]
Description: Overall survival is defined as the time from the date of randomization to the date of death. The high-risk participants whose myeloma carried del(17) subgroup was defined as the cases reported as positive for del(17) by the central laboratory combined with those cases that lacked a central laboratory result but with known del (17) by local laboratory. Participants without documentation of death at the time of the analysis were censored at the date when they were last known to be alive. Data is only reported high-risk participants with Del(17).
Time Frame: From the time of screening until disease progression and thereafter every 12 weeks until death or study termination (up to approximately 97 months)
Population: ITT population was defined as all randomized participants. Overall number analyzed is the number of participants available for analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib+ Lenalidomide + Dexamethasone | Placebo + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 36 | 33
months | 42.2 [27.56 to 56.74] | 29.4 [16.99 to 44.22]
Statistical Analysis 1: Comparison: Ixazomib+ Lenalidomide + Dexamethasone vs Placebo + Lenalidomide + Dexamethasone; Test type: Superiority; p = 0.764, Log Rank; Hazard Ratio (HR) = 0.916, 95% CI 2-sided [0.516 to 1.626] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Overall Response Rate (ORR) as Assessed by the IRC
Description: ORR was defined as the percentage of participants with Complete Response (CR) including stringent complete response (sCR), very good partial response (VGPR) and Partial Response (PR) assessed by the IRC using IMWG criteria. Percentages are rounded off to single decimal.
Time Frame: Day 1 of each cycle (every 4 weeks) until disease progression up to approximately 27 months(approximate median follow-up 15 months)
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Ixazomib+ Lenalidomide + Dexamethasone | Placebo + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 360 | 362
percentage of participants | 78.3 | 71.5

5. Secondary Outcome: Percentage of Participants With Complete Response (CR) and Very Good Partial Response (VGPR) as Assessed by the IRC
Description: Response was assessed by the IRC using International Myeloma Working Group (IMWG) Criteria. CR is defined as negative immunofixation on the serum and urine and; disappearance of any soft tissue plasmacytomas and; < 5% plasma cells in bone marrow. VGPR is defined as Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level < 100 mg per 24 hours. Percentages are rounded off to single decimal.
Time Frame: Day 1 of each cycle (every 4 weeks) until disease progression up to approximately 27 months (approximate median follow-up 15 months)
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Groups:
- Ixazomib + Lenalidomide + Dexamethasone: Ixazomib 4 mg, capsules, orally, once, on Days 1, 8 and 15; plus lenalidomide 25 mg, orally, once, on Days 1 through 21; and dexamethasone 40 mg, orally, once, on Days 1, 8, 15 and 22 of a 28-day cycle for multiple cycles until PD or unacceptable toxicity, whichever occurred first up to EOT (up to approximately 42.9 months).
Arm/Group | Ixazomib + Lenalidomide + Dexamethasone | Placebo + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 360 | 362
percentage of participants | 48.1 | 39.0

6. Secondary Outcome: Duration of Response (DOR)
Description: DOR was measured as the time in months from the date of first documentation of a confirmed response of PR or better (CR [including sCR] + PR+ VGPR) to the date of the first documented disease progression (PD) among participants who responded to the treatment. Response was assessed by the investigator using International Myeloma Working Group (IMWG) Criteria.
Time Frame: Day 1 of each cycle (every 4 weeks) until disease progression up to approximately 38 months
Population: Response-Evaluable population included all participants who received at least 1 dose of study drug, had measurable disease at baseline, and at least 1 post-baseline response assessment. Overall number analyzed is the number of participants available for analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib+ Lenalidomide + Dexamethasone | Placebo + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 281 | 252
months | 26.0 [22.51 to NA] — The upper limit of CI was not estimable due to insufficient number of participants with events. | 21.7 [17.77 to NA] — The upper limit of CI was not estimable due to insufficient number of participants with events.

7. Secondary Outcome: Time to Progression (TTP) as Assessed by the IRC
Description: TTP was measured as the time in months from the first dose of study treatment to the date of the first documented progressive disease (PD) as assessed by the IRC using IMWG criteria.
Time Frame: as for outcome 5
Population: ITT population included all randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib+ Lenalidomide + Dexamethasone | Placebo + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 360 | 362
months | 22.4 [18.73 to 27.66] | 17.6 [14.52 to 20.27]

8. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Eastern Cooperative Oncology Group (ECOG) performance score, laboratory values, vital sign measurements and reported adverse events (AEs) were collected and assessed to evaluate the safety of therapy throughout the study. An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; or congenital anomaly; or a medically important event.
Time Frame: From the date of signing of the informed consent form through 30 days after the last dose of study drug up to approximately 115 months
Population: Safety population included all randomized participants who received at least 1 dose of any study drug, regardless of their randomized treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib+ Lenalidomide + Dexamethasone | Placebo + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 361 | 359
Participants
  TEAEs | 359 | 357
  SAEs | 205 | 201

9. Secondary Outcome: Number of Participants With Change From Baseline in Pain Response
Description: Pain response was defined as 30% reduction from Baseline in Brief Pain Inventory-Short Form (BPI-SF) worst pain score over the last 24 hours without an increase in analgesic (oral morphine equivalents) use at 2 consecutive evaluations. The BPI-SF contains 15 items designed to capture the pain severity ("worst," "least," "average," and "now" [current pain]), pain location, medication to relieve the pain, and the interference of pain with various daily activities including general activity, mood, walking activity, normal work, relations with other people, sleep, and enjoyment of life. The pain severity items are rated on a 0 to 10 scale where: 0=no pain and 10=pain as bad as you can imagine and averaged for a total score of 0 (best) to 10 (Worst).
Time Frame: Baseline and end of treatment (EOT) (up to approximately 38 months)
Population: ITT population included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib+ Lenalidomide + Dexamethasone | Placebo + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 360 | 362
Participants
  Baseline | 345 | 351
  EOT | 145 | 153

10. Secondary Outcome: Change From Baseline in the European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) Questionnaire (EORTC-QLQ-C30)
Description: The EORTC-QLQ-C30 is a 30-question tool used to assess the overall quality of life in cancer participants. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact).The EORTC-QLQ-C30 Global Health Status/QOL Scale is scored between 0 and 100, where higher scores indicate better Global Health Status/QOL. Negative changes from baseline indicate deterioration in QOL or functioning and positive changes indicate improvement. Scores are linearly transformed to a 0-100 scale. High scores for the global and functional domains indicate higher quality of life or functioning. Higher scores on the symptom scales represent higher levels of symptomatology or problems.
Time Frame: Baseline, EOT and follow-up (up to approximately 97 months)
Population: ITT population included all randomized participants. Overall number analyzed is the number of participants available for analysis. Number analyzed is the number of participants available for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ixazomib+ Lenalidomide + Dexamethasone | Placebo + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 356 | 360
score on a scale
  Global Health Index: Baseline: number analyzed (Participants) | 355 | 359
  Global Health Index: Baseline | 58.4 (22.60) | 56.4 (22.12)
  Global Health Index: End of Treatment: number analyzed (Participants) | 251 | 255
  Global Health Index: End of Treatment | -6.0 (24.6) | -6.0 (23.85)
  Global Health Index: Last Follow-up: number analyzed (Participants) | 0 | 1
  Global Health Index: Last Follow-up |  | 16.7 (NA) — The SD was not estimable due to single participant with event.
  Physical Functioning: Baseline: number analyzed (Participants) | 356 | 359
  Physical Functioning: Baseline | 70.0 (21.74) | 67.3 (23.54)
  Physical Functioning: EOT: number analyzed (Participants) | 253 | 261
  Physical Functioning: EOT | -4.7 (22.61) | -6.2 (23.36)
  Physical Functioning: Last Follow-up: number analyzed (Participants) | 0 | 1
  Physical Functioning: Last Follow-up |  | 0.0 (NA) — The SD was not estimable due to single participant with event.
  Role Functioning: Baseline | 68.4 (28.75) | 64.4 (30.24)
  Role Functioning: EOT: number analyzed (Participants) | 253 | 261
  Role Functioning: EOT | -8.6 (31.27) | -8.6 (32.90)
  Role Functioning: Last Follow-up: number analyzed (Participants) | 0 | 1
  Role Functioning: Last Follow-up |  | -16.7 (NA) — The SD was not estimable due to single participant with event.
  Emotional Functioning: Baseline: number analyzed (Participants) | 355 | 360
  Emotional Functioning: Baseline | 75.1 (23.47) | 75.3 (22.22)
  Emotional Functioning: EOT: number analyzed (Participants) | 251 | 256
  Emotional Functioning: EOT | -2.1 (20.09) | -6.1 (23.16)
  Emotional Functioning: Last Follow-up: number analyzed (Participants) | 0 | 1
  Emotional Functioning: Last Follow-up |  | -25.0 (NA) — The SD was not estimable due to single participant with event.
  Cognitive Functioning: Baseline: number analyzed (Participants) | 355 | 360
  Cognitive Functioning: Baseline | 81.9 (20.42) | 81.6 (19.79)
  Cognitive Functioning: EOT: number analyzed (Participants) | 251 | 256
  Cognitive Functioning: EOT | -7.6 (20.61) | -5.8 (22.24)
  Cognitive Functioning: Last Follow-up: number analyzed (Participants) | 0 | 1
  Cognitive Functioning: Last Follow-up |  | -50.0 (NA) — The SD was not estimable due to single participant with event.
  Social Functioning: Baseline: number analyzed (Participants) | 354 | 360
  Social Functioning: Baseline | 77.9 (26.07) | 75.3 (26.47)
  Social Functioning: EOT: number analyzed (Participants) | 250 | 256
  Social Functioning: EOT | -6.9 (29.44) | -7.9 (29.37)
  Social Functioning: Last Follow-up: number analyzed (Participants) | 0 | 1
  Social Functioning: Last Follow-up |  | 0.0 (NA) — The SD was not estimable due to single participant with event.
  Fatigue: Baseline | 38.4 (23.98) | 39.5 (25.14)
  Fatigue: EOT: number analyzed (Participants) | 253 | 261
  Fatigue: EOT | 6.0 (25.38) | 6.7 (26.61)
  Fatigue: Last Follow-up: number analyzed (Participants) | 0 | 1
  Fatigue: Last Follow-up |  | 22.2 (NA) — The SD was not estimable due to single participant with event.
  Pain: Baseline | 38.0 (28.30) | 38.5 (30.99)
  Pain: EOT: number analyzed (Participants) | 253 | 261
  Pain: EOT | 2.7 (26.65) | 3.8 (30.07)
  Pain: Last Follow-up: number analyzed (Participants) | 0 | 1
  Pain: Last Follow-up |  | 0.0 (NA) — The SD was not estimable due to single participant with event.
  Nausea and Vomiting: Baseline | 5.0 (12.89) | 6.0 (13.31)
  Nausea and Vomiting: EOT: number analyzed (Participants) | 252 | 261
  Nausea and Vomiting: EOT | 3.4 (16.85) | 0.6 (19.22)
  Nausea and Vomiting: Last Follow-up: number analyzed (Participants) | 0 | 1
  Nausea and Vomiting: Last Follow-up |  | 33.3 (NA) — The SD was not estimable due to single participant with event.
  Dyspnea: Baseline | 21.2 (26.74) | 23.7 (26.68)
  Dyspnea: EOT: number analyzed (Participants) | 252 | 261
  Dyspnea: EOT | 5.7 (31.04) | 2.3 (27.33)
  Dyspnea: Last Follow-up: number analyzed (Participants) | 0 | 1
  Dyspnea: Last Follow-up |  | 0.0 (NA) — The SD was not estimable due to single participant with event.
  Insomnia: Baseline | 27.4 (31.04) | 30.5 (31.59)
  Insomnia: EOT: number analyzed (Participants) | 252 | 260
  Insomnia: EOT | 0.9 (31.41) | -0.5 (33.26)
  Insomnia: Last Follow-up: number analyzed (Participants) | 0 | 1
  Insomnia: Last Follow-up |  | 33.3 (NA) — The SD was not estimable due to single participant with event.
  Appetite Loss: Baseline | 16.9 (25.70) | 15.3 (25.21)
  Appetite Loss: EOT: number analyzed (Participants) | 253 | 260
  Appetite Loss: EOT | 4.7 (31.49) | 6.5 (28.47)
  Appetite Loss: Last Follow-up: number analyzed (Participants) | 0 | 1
  Appetite Loss: Last Follow-up |  | 0.0 (NA) — The SD was not estimable due to single participant with event.
  Constipation: Baseline: number analyzed (Participants) | 355 | 360
  Constipation: Baseline | 12.2 (22.58) | 13.5 (24.30)
  Constipation: EOT: number analyzed (Participants) | 249 | 259
  Constipation: EOT | -1.3 (26.57) | 2.2 (27.05)
  Constipation: Last Follow-up: number analyzed (Participants) | 0 | 1
  Constipation: Last Follow-up |  | 33.3 (NA) — The SD was not estimable due to single participant with event.
  Diarrhea: Baseline: number analyzed (Participants) | 355 | 360
  Diarrhea: Baseline | 6.3 (16.38) | 8.1 (18.49)
  Diarrhea: EOT: number analyzed (Participants) | 250 | 256
  Diarrhea: EOT | 17.2 (31.08) | 10.8 (31.53)
  Diarrhea: Last Follow-up: number analyzed (Participants) | 0 | 1
  Diarrhea: Last Follow-up |  | 0.0 (NA) — The SD was not estimable due to single participant with event.
  Financial Difficulties: Baseline: number analyzed (Participants) | 352 | 360
  Financial Difficulties: Baseline | 16.7 (26.15) | 18.6 (28.30)
  Financial Difficulties: EOT: number analyzed (Participants) | 250 | 256
  Financial Difficulties: EOT | 0.5 (20.69) | 1.3 (26.54)
  Financial Difficulties: Last Follow-up: number analyzed (Participants) | 0 | 1
  Financial Difficulties: Last Follow-up |  | -33.3 (NA) — The SD was not estimable due to single participant with event.

11. Secondary Outcome: Change From Baseline in the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Multiple Myeloma Module (QLQ-MY-20)
Description: The EORTC-QLQ-MY-20 is a patient-completed, 20-question quality of life questionnaire that has 4 independent subscales, 2 functional subscales (body image, future perspective), and 2 symptoms scales (disease symptoms and side-effects of treatment). The participant answers questions about their health during the past week using a 4-point scale where 1=Not at All to 4=Very Much. A negative change from Baseline indicates improvement. Scores are linearly transformed to a 0-100 scale. Higher scores on the symptom scales (e.g. Disease Symptoms, Side Effects of Treatment) represent higher levels of symptomatology or problems. High scores for Body Image and Future Perspective represent better quality of life or functioning.
Time Frame: Baseline, EOT and follow-up (up to approximately 97 months)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ixazomib+ Lenalidomide + Dexamethasone | Placebo + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 354 | 359
score on a scale
  Disease Symptoms: Baseline | 29.71 (20.850) | 30.41 (23.072)
  Disease Symptoms: EOT: number analyzed (Participants) | 248 | 255
  Disease Symptoms: EOT | -2.35 (20.752) | -2.58 (21.372)
  Disease Symptoms: Last Follow-up: number analyzed (Participants) | 1 | 0
  Disease Symptoms: Last Follow-up | 1.11 (NA) — The SD was not estimable due to single participant with event. |
  Side Effects of Treatment: Baseline | 17.23 (14.289) | 17.97 (14.682)
  Side Effects of Treatment: EOT: number analyzed (Participants) | 249 | 255
  Side Effects of Treatment: EOT | 4.52 (14.435) | 4.43 (13.955)
  Side Effects of Treatment: Last Follow-up: number analyzed (Participants) | 0 | 1
  Side Effects of Treatment: Last Follow-up |  | 37.04 (NA) — The SD was not estimable due to single participant with event.
  Body Image: Baseline: number analyzed (Participants) | 353 | 359
  Body Image: Baseline | 78.00 (29.259) | 79.48 (27.233)
  Body Image: EOT: number analyzed (Participants) | 245 | 254
  Body Image: EOT | -0.27 (29.102) | -5.38 (29.368)
  Body Image: Last Follow-up: number analyzed (Participants) | 0 | 1
  Body Image: Last Follow-up |  | -33.3 (NA) — The SD was not estimable due to single participant with event.
  Future Perspective: Baseline: number analyzed (Participants) | 353 | 359
  Future Perspective: Baseline | 56.99 (25.170) | 60.26 (25.064)
  Future Perspective: EOT: number analyzed (Participants) | 248 | 255
  Future Perspective: EOT | 2.76 (22.90) | -2.75 (22.842)
  Future Perspective: Last Follow-up: number analyzed (Participants) | 0 | 1
  Future Perspective: Last Follow-up |  | -11.11 (NA) — The SD was not estimable due to single participant with event.

12. Secondary Outcome: OS in High-Risk Participants
Description: Overall survival (OS) is defined as the time from the date of randomization to the date of death. High-risk participants are defined as participants carrying cytogenic abnormalities: del(17), translocation t(4;14), or t(14;16) as reported by the central laboratory combined with those cases that lacked a central laboratory result but with known del (17), t(4;14), or t(14;16) by local laboratory. Cytogenetic abnormalities of del(13) and +1q are not included in the analysis. Participants without documentation of death at the time of the analysis were censored at the date when they were last known to be alive. Data is only reported for high-risk participants.
Time Frame: as for outcome 3
Population: ITT population included all randomized participants. Overall number analyzed is the number of participants available for analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib+ Lenalidomide + Dexamethasone | Placebo + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 75 | 62
months | 46.9 [34.04 to 64.53] | 30.9 [24.77 to 42.25]

13. Secondary Outcome: PFS in High-Risk Participants
Description: Progression Free Survival (PFS) is defined as the time from the date of randomization to the date of first documentation of disease progression or death due to any cause, whichever occurs first. Response was assessed by independent review committee (IRC) using IMWG response criteria. High-risk participants are defined as participants carrying cytogenic abnormalities: del(17), translocation t(4;14), or t(14;16) as reported by the central laboratory combined with those cases that lacked a central laboratory result but with known del (17), t(4;14), or t(14;16) by local laboratory. Cytogenetic abnormalities of del(13) and +1q are not included in the analysis.
Time Frame: From date of randomization until disease progression or death up to approximately 38 months (approximate median follow-up 15 months)
Population: Participants from the ITT population, all randomized participants, with cytogenic abnormalities. Overall number analyzed is the number of participants available for analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib+ Lenalidomide + Dexamethasone | Placebo + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 75 | 62
months | 18.7 [13.24 to NA] — The upper limit of CI was not estimable due to insufficient number of participants with events. | 9.3 [7.36 to 15.70]

14. Secondary Outcome: Plasma Concentration Over Time for Ixazomib
Time Frame: Pre-dose and post-dose at multiple timepoints up to Cycle 10 Day 1 (each cycle length = 28 days)
Population: Safety population is defined as all subjects who received at least 1 dose of any study drug. Overall number analyzed is the number of participants available for analysis. Number analyzed is the number of participants available for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Ixazomib+ Lenalidomide + Dexamethasone | Placebo + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 335 | 5
μg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 0
  Cycle 1 Day 1 | 4.79 (NA) — The SD was not estimable due to single participant with event. |
  Cycle 1 Day 1, 1 Hour Post-Dose: number analyzed (Participants) | 330 | 4
  Cycle 1 Day 1, 1 Hour Post-Dose | 36.3 (31.3) | 0 (0)
  Cycle 1 Day 1, 4 Hours Post-Dose: number analyzed (Participants) | 321 | 4
  Cycle 1 Day 1, 4 Hours Post-Dose | 15.6 (11.1) | 0 (0)
  Cycle 1 Day 14, Pre-Dose: number analyzed (Participants) | 335 | 4
  Cycle 1 Day 14, Pre-Dose | 6.83 (10.5) | 0 (0)
  Cycle 2 Day 1, Pre-Dose: number analyzed (Participants) | 331 | 5
  Cycle 2 Day 1, Pre-Dose | 2.4 (2.4) | 0 (0)
  Cycle 2 Day 14, Pre-Dose: number analyzed (Participants) | 324 | 5
  Cycle 2 Day 14, Pre-Dose | 7.12 (8.44) | 0 (0)
  Cycle 3 Day 1, Pre-Dose: number analyzed (Participants) | 329 | 5
  Cycle 3 Day 1, Pre-Dose | 2.48 (1.69) | 0 (0)
  Cycle 4 Day 1, Pre-Dose: number analyzed (Participants) | 319 | 4
  Cycle 4 Day 1, Pre-Dose | 2.41 (1.35) | 0 (0)
  Cycle 5 Day 1, Pre-Dose: number analyzed (Participants) | 307 | 4
  Cycle 5 Day 1, Pre-Dose | 2.42 (1.49) | 0 (0)
  Cycle 6 Day 1, Pre-Dose: number analyzed (Participants) | 290 | 4
  Cycle 6 Day 1, Pre-Dose | 2.57 (3.89) | 0 (0)
  Cycle 7 Day 1, Pre-Dose: number analyzed (Participants) | 279 | 3
  Cycle 7 Day 1, Pre-Dose | 2.71 (4.79) | 0 (0)
  Cycle 8 Day 1, Pre-Dose: number analyzed (Participants) | 268 | 2
  Cycle 8 Day 1, Pre-Dose | 2.37 (1.47) | 0 (0)
  Cycle 9 Day 1, Pre-Dose: number analyzed (Participants) | 262 | 4
  Cycle 9 Day 1, Pre-Dose | 2.51 (2.13) | 0 (0)
  Cycle 10 Day 1, Pre-Dose: number analyzed (Participants) | 239 | 2
  Cycle 10 Day 1, Pre-Dose | 2.82 (5.98) | 0 (0)

15. Secondary Outcome: Overall Response Rate in Participants Defined by Polymorphism
Description: Data is reported for percentage of participants defined by polymorphism defined by polymorphisms in proteasome genes, such as polymorphism P11A in PSMB1 gene. Percentages are rounded off to single decimal.
Time Frame: as for outcome 5
Population: ITT population included all randomized participants. Overall number analyzed is the number of participants available with data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo + Lenalidomide + Dexamethasone: Ixazomib placebo-matching capsules, orally, once, on Days 1, 8 and 15; plus lenalidomide 25 mg, orally, once, on Days 1 through 21; and dexamethasone 40 mg, orally, once, on Days 1, 8, 15 and 22 of a 28-day cycle for multiple cycles until progressive disease (PD) or unacceptable toxicity, whichever occurred first up to (up to approximately 41 months).
Arm/Group | Ixazomib+ Lenalidomide + Dexamethasone | Placebo + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 117 | 115
percentage of participants | 80.3 [72.0 to 87.1] | 75.7 [66.8 to 83.2]
Statistical Analysis 1: Comparison: Ixazomib+ Lenalidomide + Dexamethasone vs Placebo + Lenalidomide + Dexamethasone; Test type: Superiority; p = 0.332, Cochran-Mantel-Haenszel — P-value is from Cochran-Mantel-Haenszel stratified by: prior therapies (1, 2 or 3), proteasome inhibitor (exposed, naïve), and ISS Stage at Screening (I or II, III); Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.69 to 2.45] — Odds ratio is from logistic regression model with prognostic factors: prior therapies (1, 2 or 3), proteasome inhibitor (exposed, naïve),and ISS Stage at Screening (I or II, III). Odds ratio > 1 favors Ixazomib

ADVERSE EVENTS:
Time Frame: From the date of signing of the informed consent form through 30 days after the last dose of study drug up to approximately 115 months
Description: The investigator had to document any occurrence of adverse events including abnormal laboratory findings. Any event spontaneously reported by the participant or observed by investigator was recorded, irrespective of the relation to study treatment. Safety population included all randomized participants who received at least 1 dose of any study drug, regardless of their randomized treatment.
Arm/Group | Ixazomib+ Lenalidomide + Dexamethasone | Placebo + Lenalidomide + Dexamethasone
All-Cause Mortality (participants affected / at risk) | 250/361 | 251/359
Serious Adverse Events (participants affected / at risk) | 205/361 | 202/359
Other Adverse Events (participants affected / at risk) | 350/361 | 342/359
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib+ Lenalidomide + Dexamethasone (N=361) | Placebo + Lenalidomide + Dexamethasone (N=359)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 5 | 6
Acute myocardial infarction (Cardiac disorders) | 1 | 2
Acute polyneuropathy (Nervous system disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute vestibular syndrome (Ear and labyrinth disorders) | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Anaemia (Blood and lymphatic system disorders) | 5 | 10
Angina pectoris (Cardiac disorders) | 2 | 3
Angina unstable (Cardiac disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0
Aortic dissection (Vascular disorders) | 0 | 1
Aortic thrombosis (Vascular disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 1
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 | 1
Asthenia (General disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Atonic urinary bladder (Renal and urinary disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 6 | 7
Atrial flutter (Cardiac disorders) | 2 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Atypical pneumonia (Infections and infestations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 8
Bacterial infection (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 1
Bartholin's cyst (Reproductive system and breast disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Bladder adenocarcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bronchitis (Infections and infestations) | 6 | 10
Bronchitis bacterial (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 2 | 3
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Campylobacter colitis (Infections and infestations) | 0 | 1
Campylobacter gastroenteritis (Infections and infestations) | 2 | 1
Candida pneumonia (Infections and infestations) | 1 | 0
Cardiac arrest (Cardiac disorders) | 3 | 3
Cardiac failure (Cardiac disorders) | 4 | 6
Cardiac failure acute (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 3
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0
Cataract (Eye disorders) | 5 | 7
Cellulitis (Infections and infestations) | 4 | 2
Central nervous system lesion (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 2
Cerebral infarction (Nervous system disorders) | 1 | 1
Cerebral small vessel ischaemic disease (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Chills (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 2 | 5
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Chronic sinusitis (Infections and infestations) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Coma (Nervous system disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 2
Complicated appendicitis (Infections and infestations) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Coronary artery thrombosis (Cardiac disorders) | 0 | 1
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Cytomegalovirus colitis (Infections and infestations) | 0 | 1
Death (General disorders) | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 5 | 7
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Dermo-hypodermitis (Infections and infestations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 12 | 3
Diarrhoea infectious (Infections and infestations) | 0 | 1
Diastolic dysfunction (Cardiac disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Endocarditis (Infections and infestations) | 0 | 1
Endocarditis staphylococcal (Infections and infestations) | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1
Enteritis infectious (Infections and infestations) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 2 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 4
Fatigue (General disorders) | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 9
Femoral hernia incarcerated (Gastrointestinal disorders) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 | 2
Femur fracture (Injury, poisoning and procedural complications) | 3 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastroenteritis (Infections and infestations) | 5 | 1
Gastroenteritis caliciviral (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 2 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 3
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 2
H1N1 influenza (Infections and infestations) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 2
Haemophilus infection (Infections and infestations) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Herpes zoster (Infections and infestations) | 3 | 3
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 4 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 3
Hyperthermia (General disorders) | 1 | 0
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 | 1
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Hypotension (Vascular disorders) | 2 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 2 | 0
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Infection (Infections and infestations) | 4 | 3
Influenza (Infections and infestations) | 8 | 5
Influenza A virus test positive (Investigations) | 1 | 2
Influenza like illness (General disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 3 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral discitis (Infections and infestations) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 3
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestine infection (Infections and infestations) | 1 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Lobular breast carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Localised infection (Infections and infestations) | 0 | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 6 | 4
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malaise (General disorders) | 2 | 1
Meningitis pneumococcal (Infections and infestations) | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Metapneumovirus infection (Infections and infestations) | 0 | 3
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Moraxella infection (Infections and infestations) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Myocardial infarction (Cardiac disorders) | 5 | 2
Myocardial ischaemia (Cardiac disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 1
Neuralgia (Nervous system disorders) | 1 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neurogenic bladder (Renal and urinary disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 2
Non-cardiac chest pain (General disorders) | 2 | 1
Oedema peripheral (General disorders) | 0 | 1
Oesophageal achalasia (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 3 | 1
Parainfluenzae virus infection (Infections and infestations) | 1 | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 5 | 4
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Penile squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Performance status decreased (General disorders) | 1 | 0
Peripheral artery aneurysm (Vascular disorders) | 1 | 0
Peripheral swelling (General disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Phlebitis superficial (Vascular disorders) | 1 | 0
Pilonidal cyst (Infections and infestations) | 0 | 1
Plasma cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Platelet count decreased (Investigations) | 3 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumococcal infection (Infections and infestations) | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 47 | 46
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonia escherichia (Infections and infestations) | 1 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0
Pneumonia haemophilus (Infections and infestations) | 2 | 0
Pneumonia influenzal (Infections and infestations) | 1 | 1
Pneumonia moraxella (Infections and infestations) | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 2
Pneumonia pseudomonal (Infections and infestations) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Postoperative wound infection (Infections and infestations) | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Proteus infection (Infections and infestations) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 2
Pseudomonas infection (Infections and infestations) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 9
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary microemboli (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Pyrexia (General disorders) | 12 | 18
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 3
Renal impairment (Renal and urinary disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory syncytial virus infection (Infections and infestations) | 1 | 2
Respiratory tract infection (Infections and infestations) | 3 | 7
Retinal vein thrombosis (Eye disorders) | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 3
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Salmonella sepsis (Infections and infestations) | 1 | 0
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Sepsis (Infections and infestations) | 4 | 5
Septic shock (Infections and infestations) | 4 | 5
Sinusitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 3
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Soft tissue inflammation (General disorders) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 5
Spinal cord compression (Nervous system disorders) | 3 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 7
Staphylococcal infection (Infections and infestations) | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0
Sudden death (General disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Syncope (Nervous system disorders) | 6 | 4
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 6
Thrombophlebitis (Vascular disorders) | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Toxic goitre (Endocrine disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Trifascicular block (Cardiac disorders) | 1 | 0
Typhoid fever (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 3
Urethral haemorrhage (Renal and urinary disorders) | 1 | 0
Urethral meatus stenosis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 2
Urinary tract infection (Infections and infestations) | 3 | 6
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 2
Vascular encephalopathy (Nervous system disorders) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Visceral leishmaniasis (Infections and infestations) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Weight decreased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib+ Lenalidomide + Dexamethasone (N=361) | Placebo + Lenalidomide + Dexamethasone (N=359)
Abdominal pain (Gastrointestinal disorders) | 37 | 36
Abdominal pain upper (Gastrointestinal disorders) | 26 | 17
Anaemia (Blood and lymphatic system disorders) | 123 | 105
Anxiety (Psychiatric disorders) | 18 | 23
Arthralgia (Musculoskeletal and connective tissue disorders) | 79 | 71
Asthenia (General disorders) | 62 | 66
Atrial fibrillation (Cardiac disorders) | 17 | 19
Back pain (Musculoskeletal and connective tissue disorders) | 97 | 82
Bone pain (Musculoskeletal and connective tissue disorders) | 33 | 34
Bronchitis (Infections and infestations) | 76 | 53
Cataract (Eye disorders) | 50 | 61
Conjunctivitis (Infections and infestations) | 34 | 10
Constipation (Gastrointestinal disorders) | 125 | 99
Contusion (Injury, poisoning and procedural complications) | 23 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 73 | 65
Decreased appetite (Metabolism and nutrition disorders) | 51 | 42
Deep vein thrombosis (Vascular disorders) | 11 | 18
Depression (Psychiatric disorders) | 19 | 18
Diarrhoea (Gastrointestinal disorders) | 186 | 153
Dizziness (Nervous system disorders) | 58 | 43
Dry eye (Eye disorders) | 22 | 6
Dry mouth (Gastrointestinal disorders) | 16 | 25
Dysgeusia (Nervous system disorders) | 23 | 15
Dyspepsia (Gastrointestinal disorders) | 33 | 31
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 7 | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 44 | 40
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 17 | 24
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 20 | 16
Erythema (Skin and subcutaneous tissue disorders) | 22 | 13
Fall (Injury, poisoning and procedural complications) | 35 | 40
Fatigue (General disorders) | 113 | 103
Gastroenteritis (Infections and infestations) | 26 | 17
Headache (Nervous system disorders) | 53 | 56
Herpes zoster (Infections and infestations) | 20 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 18 | 23
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 14 | 18
Hypertension (Vascular disorders) | 29 | 27
Hypocalcaemia (Metabolism and nutrition disorders) | 24 | 21
Hypokalaemia (Metabolism and nutrition disorders) | 60 | 51
Hypomagnesaemia (Metabolism and nutrition disorders) | 18 | 26
Influenza (Infections and infestations) | 27 | 26
Influenza like illness (General disorders) | 25 | 15
Insomnia (Psychiatric disorders) | 82 | 106
Leukopenia (Blood and lymphatic system disorders) | 28 | 19
Lower respiratory tract infection (Infections and infestations) | 16 | 18
Mood altered (Psychiatric disorders) | 12 | 21
Muscle spasms (Musculoskeletal and connective tissue disorders) | 70 | 102
Muscular weakness (Musculoskeletal and connective tissue disorders) | 21 | 28
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 33 | 39
Myalgia (Musculoskeletal and connective tissue disorders) | 22 | 16
Nasopharyngitis (Infections and infestations) | 90 | 86
Nausea (Gastrointestinal disorders) | 114 | 83
Neck pain (Musculoskeletal and connective tissue disorders) | 14 | 21
Neuropathy peripheral (Nervous system disorders) | 35 | 26
Neutropenia (Blood and lymphatic system disorders) | 112 | 99
Neutrophil count decreased (Investigations) | 26 | 28
Oedema peripheral (General disorders) | 97 | 76
Oral candidiasis (Infections and infestations) | 17 | 19
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 | 21
Pain in extremity (Musculoskeletal and connective tissue disorders) | 54 | 41
Paraesthesia (Nervous system disorders) | 33 | 19
Peripheral sensory neuropathy (Nervous system disorders) | 88 | 61
Peripheral swelling (General disorders) | 20 | 7
Pharyngitis (Infections and infestations) | 16 | 22
Platelet count decreased (Investigations) | 36 | 22
Pneumonia (Infections and infestations) | 46 | 33
Pruritus (Skin and subcutaneous tissue disorders) | 45 | 32
Pyrexia (General disorders) | 55 | 71
Rash (Skin and subcutaneous tissue disorders) | 20 | 11
Rash macular (Skin and subcutaneous tissue disorders) | 26 | 29
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 34 | 15
Respiratory tract infection (Infections and infestations) | 23 | 30
Sinusitis (Infections and infestations) | 25 | 21
Thrombocytopenia (Blood and lymphatic system disorders) | 95 | 44
Tremor (Nervous system disorders) | 22 | 38
Upper respiratory tract infection (Infections and infestations) | 97 | 83
Urinary tract infection (Infections and infestations) | 43 | 34
Vision blurred (Eye disorders) | 26 | 18
Vomiting (Gastrointestinal disorders) | 93 | 47
Weight decreased (Investigations) | 36 | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.

DOCUMENTS (2):
  • Study Protocol (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/37/NCT01564537/Prot_000.pdf
  • Statistical Analysis Plan (2014-12-16): https://cdn.clinicaltrials.gov/large-docs/37/NCT01564537/SAP_001.pdf